CLINICAL TRIAL: NCT04584866
Title: Semi-sitting Versus Supine Position in Endoscopic Skull Base Surgery (PosESS-Study) - Study Protocol for a Randomized-controlled Single-blinded Superiority Trial
Brief Title: Semi-sitting Versus Supine Position in Endoscopic Skull Base Surgery
Acronym: PosESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-02115; ch20Rychen
Record Dates: First submitted 2020-10-05; First posted 2020-10-14 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Pituitary Adenoma
Keywords: endoscopic endonasal pituitary surgery; endoscopic skull base surgery; intracranial venous pressure; venous air embolism
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Supine Position

STUDY DESIGN:
Intervention Model Description: prospective randomized single-blinded controlled superiority trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Intervention (Active Comparator): Endonasal endoscopic pituitary surgery in semi-sitting position
  Interventions: Procedure: Endonasal endoscopic pituitary surgery in semi-sitting position
- Control Intervention (Active Comparator): Endonasal endoscopic pituitary surgery in supine position
  Interventions: Procedure: Endonasal endoscopic pituitary surgery in supine position

INTERVENTIONS:
Procedure: Endonasal endoscopic pituitary surgery in semi-sitting position — Patients will be placed in semi-sitting position. To achieve the semi-sitting position, the patient is placed in supine position. The operating table is then separated and flexed to elevate the torso (angle of 30°). The head, which is fixed in a head clamp, is slightly flexed to bring the floor of the sella right in front of the surgeon and gently rotated toward the operating team.
  Arms: Study Intervention
Procedure: Endonasal endoscopic pituitary surgery in supine position — Patients will be operated in the standard supine neutral position
  Arms: Control Intervention

SUMMARY:
This study is to prospectively compare the standard supine (control group) and the semi-sitting position (head elevation of 30°; intervention group) in endoscopic endonasal pituitary surgery.

DETAILED DESCRIPTION:
The endonasal endoscopic approach (EEA) for pituitary surgery is standardly performed with the patient in supine position (SP). The semi-sitting position (SSP) is routinely used for the traditional microscopic transsphenoidal approach and also for posterior fossa surgery. The SSP results in lower intracranial pressure when compared to the supine position due to decreased venous congestion. As a result, intraoperative bleeding may be reduced, potentially leading to decreased surgical morbidity and improved surgical workflow. Studies during endoscopic sinus surgery have shown a significant reduction of blood loss when the patient is placed in a reverse Trendelenburg position with a head elevation of 30°. This study is to prospectively compare the standard supine (control group) and the semi-sitting position (head elevation of 30°; intervention group) in endoscopic endonasal pituitary surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a presumed pituitary pathologies who are suitable for endoscopic endonasal surgical resection

Exclusion Criteria:

* Patients with known hemorrhagic or thrombophilic disorders
* Patients with conditions associated with high central venous pressure: congestive heart failure, pulmonary hypertension, chronic obstructive pulmonary disease (COPD), interstitial lung disease, pregnancy
* Patients with poor cardiopulmonary condition (unable to perform 4 metabolic equivalents without stopping (climb a flight of stairs))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss | Intraoperative
  Intraoperative blood loss, calculated as follow: volume in the suction bag minus volume of rinsing water in Milliliters (ml). The surgery is divided into four steps: 1. endonasal phase, 2. osteodural exposure. 3. sellar stage and 4. skull base defect closure. For each step, the primary outcome will be assessed.
Frequency of interruption of the surgical workflow due to disturbing blood or a bleeding in the surgical field (number) | During surgery
  Frequency of interruption of the surgical workflow due to disturbing blood or a bleeding in the surgical field. This will be assessed by an independent blinded neurosurgeon, who will watch the operative video after the surgery.

SECONDARY OUTCOMES:
Change in intraoperative Mean Arterial Pressure (MAP) | Intraoperative
  MAP will be monitored during the whole surgery using the software Copra ©, which allows a continuous data extraction
Amount of intravenous fluid administered during surgery (ml) | Intraoperative
  Amount of intravenous fluid administered during surgery (ml)
Need for vasoactive drugs (vasopressors) (number) | at Day 1 (day of surgery)
  Need for vasoactive drugs (vasopressors) (number)
Incidence of air embolism (number) | at Day 1 (day of surgery)
  Incidence of air embolism (number)
Operative time (minutes) | During surgery
  Operative time (minutes)
Degree of descent or prolapse of the diaphragma sellae into the sellar cavity | Intraoperative
  Intraoperative assessment of the degree of descent or prolapse of the diaphragma sellae into the sellar cavity (class I to V, according to the classification of Abdelmaksoud et al)
Occurrence of a cerebrospinal fluid (CSF) leak during surgery (assessed by the operating neurosurgeon) (yes/ no) | During surgery
  Occurrence of a cerebrospinal fluid (CSF) leak during surgery (assessed by the operating neurosurgeon)
Surgical ergonomics | at Day 1 (day of surgery)
  Surgical ergonomics assessed by the means of a standardized questionnaire. The surgeon will be asked to rate the intensity of neck and arm discomfort and the frequency of surgical flow interruption due to a suboptimal trajectory of the endoscope and the instruments due to the patient Position (1 = no discomfort, 2 = medium discomfort, 3 = high discomfort).
Incidence of rhinoliquorrhoea (number) | at 3 months after surgery
  Incidence of rhinoliquorrhoea (number)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rychen, Principal Investigator — Department of Neurosurgery, University Hospital Basel
Locations (1):
- Department of Neurosurgery, University Hospital Basel, Basel, Switzerland